CLINICAL TRIAL: NCT06325826
Title: The Study of the Validation of General Evaluation Score (GES) in the Prediction of Hepatocellular Carcinoma Risk Among Patients With Advanced Fibrosis and Cirrhosis Who Achieved Sustained Virological Response for Hepatitis C Virus After Direct Acting Antiviral Drugs
Status: Active, not recruiting | Type: Observational
Sponsor: Egyptian Liver Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: GES
Record Dates: First submitted 2024-03-16; First posted 2024-03-22 (Actual); Last update posted 2024-03-26 (Actual); Status verified 2024-03

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Group 1
  Interventions: Diagnostic Test: General Evaluation Score (GES)

INTERVENTIONS:
Diagnostic Test: General Evaluation Score (GES) — According to Evaluation of GES scores Patient will be classified into three groups based on GES score low risk group (score ≤6 points), intermediate risk group (score 6-7.5 points), and high-risk group (score >7.5 points)

SUMMARY:
This cohort study aims to evaluate the validation of general evaluation score in the prediction of hepatocellular carcinoma risk among patients with advanced fibrosis (F3) and cirrhosis (F4) who achieved sustained virological response for hepatitis c virus after direct acting antiviral drugs and determine the group of these patients who require intensified surveillance.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients aged 18 years or older.
* Patients with compensated advanced chronic liver disease (cACLD) according to Baveno VI consensus (F3-F4)
* achieved SVR for HCV after DAAs.

Exclusion Criteria:

* Previous interferon (IFN) treatment.
* Hepatitis B virus (HBV) or human immune-deficiency virus (HIV) co-infection.
* Current hepatocellular carcinoma (HCC) or other malignancies.
* Previous history of HCC or HCC intervention.
* Liver cell failure, liver transplantation or renal impairment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with advanced fibrosis (F3) and cirrhosis (F4) who achieved SVR for HCV after DAAs
Sampling Method: Non-Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Hepatocellular Carcinoma | 24 month
  Number of Participants develop New Hepatocellular Carcinoma

CONTACTS AND LOCATIONS:
Locations (1):
- Egyptian Liver Hospital, Ţalkhā, Dakahlia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided